CLINICAL TRIAL: NCT00192790
Title: Clinical and Experimental Pain Perception is Attenuated in Patients With Painless Myocardial Infarction
Brief Title: Pain Perception is Attenuated in Patients With Painless Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Other Study IDs: ZSA1871CTIL
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Myocardial Infarction; Myocardial Ischemia
Keywords: Therma,pain, Silent myocardial ischemia, catastrophizing
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To explore whether reduced systemic pain perception in response to painful stimuli and personality pain related variables characterizes silent MI patients.

DETAILED DESCRIPTION:
Objective: Silent myocardial infarction (MI) is an event of severe myocardial ischemia without pain experience. The lack of pain alarm leads to increased morbidity and mortality, because the patients do not sick timely medical treatment. This study aims to explore whether reduced systemic pain perception in response to painful stimuli and personality pain related variables characterizes silent MI patients.

Methods: Level of chest pain intensity was assessed by visual analogue scale (VAS), range from 0 (no pain) to 100 (maximal pain). Heat pain threshold, magnitude estimation of supra-threshold painful stimuli at 47ºC as well as pain catastrophizing scores were assessed in 90 acute MI patients (mean age 66±12.1, range 33-79) with chest pain (n=65) and without pain symptoms(n=25). All stimuli were performed by Thermal Sensory Analysis (TSA) and applied to the right forearm.

Results: The demographic variables, history of ischemic heart, risk factors for coronary artery disease, ST-T segment changes on ECG and troponin levels were similar in both groups. Greater intensity of chest pain VAS scores was inversely correlated with lower pain threshold (r= -0.417, p<0.001), and directly associated with higher pain scores in response to the heat pain (r=0.354, p=0.002). Patients with painful MI demonstrated lower pain threshold (41.9±3.6 vs. 44.9±3.8, p=0.001), higher VAS scores in response to the supra-threshold painful stimuli (50.2 ±21.8 vs. 27.0±25.2, p=0.002), and higher catastrophizing level (10.6±12.0 vs. 5.4±8.8, p=0.032). Chest pain complaint was not related to ST-T changes as well as concomitant diseases.

Conclusions: This study suggests that reduced systemic pain perception as well as cognitive personality variables play an important role in the etiology of Silent MI.

ELIGIBILITY:
Inclusion Criteria:All patients with painless or painful myocardial infarction -

Exclusion Criteria:Patients who can't give informed concent or couldn't cooperate

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-01; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaher S. Azzam, MD, Principal Investigator — Rambam Medical Center, The Ruth & Bruce Rappaport Faculty of Medicine Technion
Locations (1):
- RAMBAM Health Care Campus, Internal Medicine "B" & Cardiology, Haifa, Israel

REFERENCES:
- [Derived] Granot M, Khoury R, Berger G, Krivoy N, Braun E, Aronson D, Azzam ZS. Clinical and experimental pain perception is attenuated in patients with painless myocardial infarction. Pain. 2007 Dec 15;133(1-3):120-7. doi: 10.1016/j.pain.2007.03.017. Epub 2007 Apr 25. PMID 17462825